CLINICAL TRIAL: NCT01350856
Title: A Multicentre, Randomised Trial to Detect in Vivo Resistance of Plasmodium Falciparum to Artesunate in Patients With Uncomplicated Malaria.
Brief Title: Tracking Resistance to Artemisinin (TRAC)
Acronym: TRAC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Mahidol University (Other); Worldwide Antimalarial Resistance Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BAKMAL1101
Record Dates: First submitted 2011-04-19; First posted 2011-05-10 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Falciparum Malaria
Keywords: Uncomplicated P. falciparum malaria
MeSH Terms: conditions — Malaria, Falciparum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Artesunate 2 (Active Comparator): Artesunate 2 mg/kg/day for 3 days followed by a full course of either artemether-lumefantrine or DHA-piperaquine or artesunate-mefloquine or artesunate-amodiaquine
  Interventions: Drug: Artesunate 2
- Artesunate 4 (Experimental): Artesunate 4 mg/kg/day for 3 days followed by a full course of either artemether-lumefantrine or DHA-piperaquine or artesunate-mefloquine or artesunate-amodiaquine
  Interventions: Drug: Artesunate 4

INTERVENTIONS:
Drug: Artesunate 2 — Artesunate 2 mg/kg/day for 3 days followed by a full course of either artemether-lumefantrine or DHA-piperaquine or artesunate-mefloquine or artesunate-amodiaquine
  Arms: Artesunate 2
Drug: Artesunate 4 — Artesunate 4 mg/kg/day for 3 days followed by a full course of either artemether-lumefantrine or DHA-piperaquine or artesunate-mefloquine or artesunate-amodiaquine
  Arms: Artesunate 4

SUMMARY:
Because the artemisinins are the most potent antimalarial drugs, the reduction in parasite numbers is rapid. Therefore, early measures of reducing parasite counts are needed. This study will look at conventional markers of parasite reduction e.g. parasite clearance time, parasite reduction ratio, and the time to achieve a fall of 50%, 90% and 99% of the pre-treatment parasitaemia.

Defining artemisinin resistance requires the use of artesunate (AS) alone because it is now appreciated that the partner drug in a combination treatment has a significant impact on the rate of parasite clearance. This study will dose patients for 3 days with AS alone (or longer until parasites clear) and measure the parasite count frequently in order to be able to define an accurate regression line of a graph of the natural logarithm of the parasite count (Y axis) versus time (X axis). This will be followed by a full course of an artemisinin combination therapy (ACT). Two different dose regimens of artesunate will be compared at all sites except those in western Cambodia, as unpublished observations from the Thai-Myanmar border suggest the standard lower daily dose of 2mg/kg may enable the earlier detection of low level resistance than a 4mg/kg daily dose.

DETAILED DESCRIPTION:
Background:

Artemisinins are the cornerstone of current antimalarial treatment. Evidence of reduced susceptibility to artemisinins in Western Cambodia was first presented in January 2007 and confirmed in a subsequent detailed pharmacokinetic-pharmacodynamic study conducted by our group. Artemisinin resistance was manifest by a marked slowing of parasite clearance. The spread of highly artemisinin resistant falciparum malaria would have devastating consequences for malaria control and elimination. The response to artemisinin resistance in P. falciparum depends critically upon answering one pivotal question: how far has it spread? This research proposal focuses on filling critical gaps in knowledge that are essential to planning an effective response.

Objectives/Hypothesis/Questions:

This is a multi-centre study with the primary objective of comparing the P. falciparum parasite clearance compared to a reference parasite clearance rate obtained from historical data in artemisinin sensitive falciparum malaria.

The aim of this large scale study is to determine if artemisinin resistance has spread and if so, how far it has spread.

Research design:

This is a multi-centre, open-label randomised trial to assess the clearance rates of peripheral blood P. falciparum parasitaemias in patients with acute uncomplicated falciparum malaria treated with two different doses of artesunate.

The study will recruit patients with acute uncomplicated P. falciparum malaria. The total number of patients for this study is expected to be 1800.

Patients will be randomised 1:1 to receive either:

* AS2: Artesunate 2 mg/kg/day for 3 days OR
* AS4: Artesunate 4 mg/kg/day for 3 days
* followed by a full course of Artesunate- mefloquine (MAS3) Patients will be hospitalised for at least the 1st three days. During hospitalisation, patients will have malaria parasite count done at 0, 4, 6, 8, 12, then every 6 hours until parasite clearance. The weekly follow up is until day 14 (on Day 7 and Day 14).

Value and significance of the research The study aims to address a simple but crucial question regarding artemisinin resistance for which currently there is no answer: has artemisinin resistant Plasmodium falciparum spread from Western Cambodia? The results will determine how to approach the subsequent efforts; strengthening of strategies for eliminating the resistant parasites in Western Cambodia if the resistance is confined to this area, or for containment and malaria control if the resistant parasites have already spread.

Potential outcomes Within one year we expect to produce a map of the geographical extent, prevalence and severity of artemisinin resistance.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged from 6 months to 65 years old, inclusive
* Acute uncomplicated P. falciparum malaria, confirmed by positive blood smear with asexual forms of P. falciparum (or mixed with non-falciparum species)
* Asexual P. falciparum parasitaemia: 10,000 to 200,000/uL, determined on a thin or thick blood film
* Fever defined as > 37.5°C tympanic temperature or a history of fever within the last 24 hours
* Written informed consent (by legally acceptable representative in case of children)
* Willingness and ability of the patients/guardians to comply with the study protocol for the duration of the study

Exclusion Criteria:

* Signs of severe/complicated malaria (WHO, 2000)
* Haematocrit < 25% or haemoglobin (Hb) < 8 g/dL at enrollment
* Acute illness other than malaria requiring treatment
* For females: pregnancy, breast feeding
* Patients who have received artemisinin or a derivative or an artemisinin-containing combination therapy (ACT) within the previous 7 days
* History of allergy or known contraindication to artemisinins, or to the ACT to be used at the site
* Previous splenectomy

Ages: 6 Months to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1700 (Actual)
Dates: Start 2011-05; Primary Completion 2014-04 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Parasite clearance rate | Day 42
  Defined by the slope of the linear portion of the natural logarithm parasite clearance curve.

SECONDARY OUTCOMES:
Parasite clearance time | Day 42
  Assessed by microscopy
Parasite reduction rates and ratios | Day 42
  Assessed by microscopy and quantitative PCR.
Time for parasite count to fall | 50%, 90%, and 99%
  Time for parasite count to fall to 50%, 90%, and 99% of initial parasite density
Fever clearance time | > 24 hours
  The time taken for tympanic temperature to fall below 37˚C and remain there for at least 24 hours
Gametocytemia in patients | days 0, 3, 7 and 14
  Proportion of patients with gametocytemia before, during and after treatment with artesunate, assessed at admission, on days 3, 7 and 14, stratified by presence of gametocytes at enrolment
Gametocyte carriage rates | 14 days
In vitro susceptibility of P.falciparum to artemisinins | Day 42
  Measure the inhibitory concentrations (IC) 50, IC90, IC99 of P. falciparum responses to artemisinins ex vivo
Pharmacokinetics relationships for artesunate and Dihydroartemisinin (DHA) | Day 42
  Measure half-life, Cmax, AUC, Tmax of artesunate and DHA.
Parasite molecular markers of drug resistance | Day 42
  To identify the parasite specific molecular marker which is correlated to artemisinin resistance
Identification of host factors that correlate with slow parasite clearance | Day 42
  To identify host factors influencing the clearance of P. falciparum, e.g. haemoglobinopathies and G6PD deficiency
Efficacy at D42 | Day 42
  The cure rate of artesunate plus ACT treatments at 42 day of follow up.
Pharmacodynamics relationships for artesunate and Dihydroartemisinin (DHA) | Day 42

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas J White, DSc MD, Principal Investigator — Mahidol Oxford Tropical Medicine Research Unit
Locations (19):
- Ramu Upazila Health Complex, Cox's Bazaar, Bangladesh
- Burma (5):
  - Myitkyina, Myitkyina, Kachin State
  - Day Bu Noh, Luthaw, Kayin State
  - Pyin Oo Lwin, Mandalay, Mandalay Region
  - Thabeikkyin Hospital, Thabeikkyin, Mandalay Region
  - Shwe Kyin Hospital, Shwe Kyin
- Cambodia (4):
  - Pursat Referral Hospital, Pursat, Pursat
  - Pailin General Hospital, Pailin
  - District Referral Hospital, Preah Vihear
  - District Referral Hospital, Rattanakiri
- Kingasani Health Centre, Kinshasa, Democratic Republic of the Congo
- Sulkapara Block Primary Health Center, West Bengal, West Bengal, India
- Pingilikani Dispensary, Kilifi, Kenya
- Phouvong District Hospital, Phouvong, Attapeu, Laos
- University of Ilorin Teaching Hospital, Ilorin, Nigeria
- Thailand (3):
  - Shoklo Malaria Research Unit, Mae Sot, Changwat Tak
  - Kraburi Hospital, Ranong
  - Phusing Hospital, Si Sa Ket
- Phuoc Long Hospital, Bình Phước, Binh Phuoc, Vietnam

REFERENCES:
- [Derived] Ashley EA, Dhorda M, Fairhurst RM, Amaratunga C, Lim P, Suon S, Sreng S, Anderson JM, Mao S, Sam B, Sopha C, Chuor CM, Nguon C, Sovannaroth S, Pukrittayakamee S, Jittamala P, Chotivanich K, Chutasmit K, Suchatsoonthorn C, Runcharoen R, Hien TT, Thuy-Nhien NT, Thanh NV, Phu NH, Htut Y, Han KT, Aye KH, Mokuolu OA, Olaosebikan RR, Folaranmi OO, Mayxay M, Khanthavong M, Hongvanthong B, Newton PN, Onyamboko MA, Fanello CI, Tshefu AK, Mishra N, Valecha N, Phyo AP, Nosten F, Yi P, Tripura R, Borrmann S, Bashraheil M, Peshu J, Faiz MA, Ghose A, Hossain MA, Samad R, Rahman MR, Hasan MM, Islam A, Miotto O, Amato R, MacInnis B, Stalker J, Kwiatkowski DP, Bozdech Z, Jeeyapant A, Cheah PY, Sakulthaew T, Chalk J, Intharabut B, Silamut K, Lee SJ, Vihokhern B, Kunasol C, Imwong M, Tarning J, Taylor WJ, Yeung S, Woodrow CJ, Flegg JA, Das D, Smith J, Venkatesan M, Plowe CV, Stepniewska K, Guerin PJ, Dondorp AM, Day NP, White NJ; Tracking Resistance to Artemisinin Collaboration (TRAC). Spread of artemisinin resistance in Plasmodium falciparum malaria. N Engl J Med. 2014 Jul 31;371(5):411-23. doi: 10.1056/NEJMoa1314981. PMID 25075834